CLINICAL TRIAL: NCT02780609
Title: Phase 1/2 Investigator Sponsored Study of Selinexor in Combination With High-Dose Melphalan Before Autologous Hematopoietic Cell Transplantation for Multiple Myeloma
Brief Title: Selinexor Plus High-Dose Melphalan (HDM) Before Autologous Hematopoietic Cell Transplantation for Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18630
Record Dates: First submitted 2016-05-20; First posted 2016-05-23 (Estimated); Results first posted 2022-05-03 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Multiple Myeloma
Keywords: autologous hematopoietic cell transplantation (HCT); high-dose melphalan; selinexor
MeSH Terms: conditions — Multiple Myeloma | interventions — selinexor; Melphalan; Dexamethasone; Calcium Dobesilate; fosaprepitant; Antiemetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Selinexor Plus HDM HCT (Experimental): The conditioning regimen begins 3 days prior to autologous transplant. Day 0 is the day of the autologous hematopoietic cell transplant. Melphalan will be given intravenously (IV) on Day -3 and Day -2; Dexamethasone will be given through via IV on Day -3, Day -2 and Day -1; fosaprepitant at 150 IV on days -3 and -2 will be given to patients an an antiemetic.Selinexor will be taken by mouth (PO) daily on the same day participants receive chemotherapy with melphalan.
  Interventions: Drug: Selinexor; Drug: Melphalan; Drug: Dexamethasone; Procedure: Autologous Hematopoietic Cell Transplantation (HCT); Drug: Fosaprepitant

INTERVENTIONS:
Drug: Selinexor — Selinexor will be given orally 2 to 3 hours prior to high dose-melphalan IV infusion. Phase I: Dose escalation beginning with 40 mg to determine the recommended Phase II dose (RPh2D). Phase II: Treatment at RPh2D.
  Other Names: KPT-330
Drug: Melphalan — Melphalan 100 mg/m^2 IV over 30-45 minutes.
  Other Names: Alkeran
Drug: Dexamethasone — Dexamethasone 20 mg PO (or IV) daily (on days -3, -2 and -1).
  Other Names: Decadron
Procedure: Autologous Hematopoietic Cell Transplantation (HCT) — Participant's own stem cells are collected from their blood, frozen, then given back to them after chemotherapy.
Drug: Fosaprepitant — Fosaprepitant at 150 mg IV on days -3 and -2.
  Other Names: antiemetic agent; Standare of Care

SUMMARY:
Phase I: The primary purpose of this study phase is to determine the best dose also referred to as the maximum tolerated dose (MTD) of Selinexor when used in combination with high-dose melphalan as a conditioning regimen for hematopoietic cell transplant.

Phase II: The primary purpose of this study phase is to assess the complete response (CR) conversion rate.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older with histologically confirmed multiple myeloma
* Achieving partial response (PR) or very good partial response (VGPR) with systemic chemotherapy
* Received less than 4 lines of anti-myeloma therapy.
* Karnofsky performance status of >= 70%
* Adequate pulmonary, cardiac, hepatic and renal function as outlined in the protocol
* Signed informed consent form in accordance with institutional policies prior to the initiation of high-dose therapy

Exclusion Criteria:

* Non-secretory multiple myeloma
* Have achieved complete response (CR) prior to autologous hematopoietic cell transplantation (HCT)
* Central nervous system (CNS) involvement
* Uncontrolled bacterial, viral or fungal infections
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Prior malignancies within the last 5 years except resected basal cell carcinoma or treated cervical carcinoma in situ.
* Females who are pregnant or breastfeeding
* Have received other investigational drugs within 14 days prior to screening
* Prior autologous or allogeneic HCT
* Prior organ transplant or autoimmune disease requiring immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taiga Nishihori, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Turner JG, Cui Y, Bauer AA, Dawson JL, Gomez JA, Kim J, Cubitt CL, Nishihori T, Dalton WS, Sullivan DM. Melphalan and Exportin 1 Inhibitors Exert Synergistic Antitumor Effects in Preclinical Models of Human Multiple Myeloma. Cancer Res. 2020 Dec 1;80(23):5344-5354. doi: 10.1158/0008-5472.CAN-19-0677. Epub 2020 Oct 6. PMID 33023948
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 Level 1: Selinexor Plus HDM HCT: 40 mg Selinexor given orally 2 to 3 hours prior to high dose-melphalan IV infusion Melphalan: Melphalan 100 mg/m^2 IV over 30-45 minutes. Dexamethasone: Dexamethasone 20 mg PO (or IV) daily (on days -3, -2 and -1). Autologous Hematopoietic Cell Transplantation (HCT): Participant's own stem cells are collected from their blood, frozen, then given back to them after chemotherapy.
  Fosaprepitant: Fosaprepitant at 150 mg IV on days -3 and -2.
- Phase 1 Level 2: Selinexor Plus HDM HCT: 60 mg Selinexor given orally 2 to 3 hours prior to high dose-melphalan IV infusion Melphalan: Melphalan 100 mg/m^2 IV over 30-45 minutes. Dexamethasone: Dexamethasone 20 mg PO (or IV) daily (on days -3, -2 and -1). Autologous Hematopoietic Cell Transplantation (HCT): Participant's own stem cells are collected from their blood, frozen, then given back to them after chemotherapy.
  Fosaprepitant: Fosaprepitant at 150 mg IV on days -3 and -2.
- Phase 1 Level 3: Selinexor Plus HDM HCT; Phase 2: Selinexor Plus HDM HCT: 80 mg Selinexor given orally 2 to 3 hours prior to high dose-melphalan IV infusion Melphalan: Melphalan 100 mg/m^2 IV over 30-45 minutes. Dexamethasone: Dexamethasone 20 mg PO (or IV) daily (on days -3, -2 and -1). Autologous Hematopoietic Cell Transplantation (HCT): Participant's own stem cells are collected from their blood, frozen, then given back to them after chemotherapy.
  Fosaprepitant: Fosaprepitant at 150 mg IV on days -3 and -2.
Period: Overall Study
Arm/Group | Phase 1 Level 1: Selinexor Plus HDM HCT | Phase 1 Level 2: Selinexor Plus HDM HCT | Phase 1 Level 3: Selinexor Plus HDM HCT | Phase 2: Selinexor Plus HDM HCT
Started | 3 | 3 | 6 | 10
Completed | 3 | 3 | 6 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 Level 1: Selinexor Plus HDM HCT | Phase 1 Level 2: Selinexor Plus HDM HCT | Phase 1 Level 3: Selinexor Plus HDM HCT | Phase 2: Selinexor Plus HDM HCT | Total
Number analyzed (Participants) | 3 | 3 | 6 | 10 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5 | 9 | 19
  >=65 years | 0 | 1 | 1 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 4 | 9
  Male | 2 | 2 | 3 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6 | 10 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 3 | 5
  White | 3 | 2 | 5 | 7 | 17
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Recommended Phase II Dose (RPh2D)
Description: RPh2D/Maximum Tolerated Dose (MTD) of Selinexor when used in combination with high-dose melphalan as a conditioning regimen for hematopoietic cell transplant. MTD: the highest dose level at which 1 or less of 6 participants experience a dose limiting toxicity (DLT).
Time Frame: Up to 3 months
Measure: Number; unit: mg
Arm/Group | Selinexor Plus HDM HCT
Number analyzed (Participants) | 12
mg | 80

2. Primary Outcome: Complete Response (CR)
Description: Complete response (CR) conversion rate. CR: Negative immunofixation of serum and urine, disappearance of any soft tissue plasmacytomas, and ≤ 5% plasma cells in bone marrow.
  tissue plasmacytomas, and ≤ 5% plasma cells in bone marrow.
  Complete Response conversion rate. CR: Negative immunofixation of serum and urine, disappearance of any soft tissue plasmacytomas, and ≤ 5% plasma cells in bone marrow.
Time Frame: 3 months post HCT
Measure: Number; unit: percentage of participants with CR
Groups:
- Phase 1 Level 2: Selinexor Plus HDM HCT: 60 mg Selinexor given orally 2 to 3 hours prior to high dose-melphalan IV infusion
  Melphalan: Melphalan 100 mg/m^2 IV over 30-45 minutes.
  Dexamethasone: Dexamethasone 20 mg PO (or IV) daily (on days -3, -2 and -1).
- Phase 1 Level 3: Selinexor Plus HDM HCT: 80 mg Selinexor given orally 2 to 3 hours prior to high dose-melphalan IV infusion
  Melphalan: Melphalan 100 mg/m^2 IV over 30-45 minutes.
  Dexamethasone: Dexamethasone 20 mg PO (or IV) daily (on days -3, -2 and -1).
Arm/Group | Phase 1 Level 1: Selinexor Plus HDM HCT | Phase 1 Level 2: Selinexor Plus HDM HCT | Phase 1 Level 3: Selinexor Plus HDM HCT | Phase 2: Selinexor Plus HDM HCT
Number analyzed (Participants) | 3 | 3 | 6 | 10
percentage of participants with CR | 0 | 33.3 | 16.6 | 10

3. Other Pre Specified Outcome: Phase 1 and Phase 2 Percentage of Participants Treated at Dose Level 3/RP2D With Progression Free Survival (PFS)
Description: Progression Free Survival defined as the time from start of treatment to the time of progression or death.
Time Frame: at 24 months
Population: All evaluable participants treated at dose level 3/RP2D.
Measure: Number (95% Confidence Interval); unit: percent of participants
Groups:
- Phase 1 Dose Level 3 and Phase 2: Selinexor Plus HDM HCT: 80 mg Selinexor given orally 2 to 3 hours prior to high dose-melphalan IV infusion
  Melphalan: Melphalan 100 mg/m^2 IV over 30-45 minutes.
  Dexamethasone: Dexamethasone 20 mg PO (or IV) daily (on days -3, -2 and -1).
  Autologous Hematopoietic Cell Transplantation (HCT): Participant's own stem cells are collected from their blood, frozen, then given back to them after chemotherapy.
  Fosaprepitant: Fosaprepitant at 150 mg IV on days -3 and -2.
Arm/Group | Phase 1 Dose Level 3 and Phase 2: Selinexor Plus HDM HCT
Number analyzed (Participants) | 15
percent of participants | 66.7 [35.8 to 85.4]

4. Other Pre Specified Outcome: Overall Survival (OS)
Description: Rate of participants' survival at time of evaluation.
Time Frame: at 24 months
Population: All evaluable participants treated at dose level 3/RP2D.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Phase 1 Dose Level 3 and Phase 2: Selinexor Plus HDM HCT
Number analyzed (Participants) | 15
percent | 95.2 [70.7 to 99.3]

5. Other Pre Specified Outcome: Rate of Minimal Residual Disease (MRD)
Description: Rate of participants who did not have Minimal Residual Disease (MRD) as assessed by flow cytometry.
Time Frame: 3 months post HCT
Population: Evaluable participants
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1 Level 1: Selinexor Plus HDM HCT | Phase 1 Level 2: Selinexor Plus HDM HCT | Phase 1 Level 3: Selinexor Plus HDM HCT | Phase 2: Selinexor Plus HDM HCT
Number analyzed (Participants) | 3 | 2 | 6 | 9
percentage of participants | 33.3 | 100 | 16.7 | 33.3

ADVERSE EVENTS:
Time Frame: Adverse events collected from date on study to 30 days after last treatment date, a total of 3 years and 8 months.
Arm/Group | Phase 1 Level 1: Selinexor Plus HDM HCT | Phase 1 Level 2: Selinexor Plus HDM HCT | Phase 1 Level 3: Selinexor Plus HDM HCT | Phase 2: Selinexor Plus HDM HCT
All-Cause Mortality (participants affected / at risk) | 2/3 | 0/3 | 2/6 | 0/10
Serious Adverse Events (participants affected / at risk) | 3/3 | 2/3 | 3/6 | 5/10
Other Adverse Events (participants affected / at risk) | 3/3 | 2/3 | 6/6 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Level 1: Selinexor Plus HDM HCT (N=3) | Phase 1 Level 2: Selinexor Plus HDM HCT (N=3) | Phase 1 Level 3: Selinexor Plus HDM HCT (N=6) | Phase 2: Selinexor Plus HDM HCT (N=10)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 5 (5)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck edema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Level 1: Selinexor Plus HDM HCT (N=3) | Phase 1 Level 2: Selinexor Plus HDM HCT (N=3) | Phase 1 Level 3: Selinexor Plus HDM HCT (N=6) | Phase 2: Selinexor Plus HDM HCT (N=10)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (8)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2) | 5 (5)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 8 (17)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 10 (27)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 10 (28)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Abdominal infection
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-06): https://cdn.clinicaltrials.gov/large-docs/09/NCT02780609/Prot_SAP_000.pdf